CLINICAL TRIAL: NCT06438718
Title: Spanish Language Validation, Validity and Reliability Testing of Frail´BESTest in Frail Institutionalized Residents Over 60 Years of Age With Mild Cognitive Impairment
Brief Title: Spanish Linguistic Validation, Validity and Reliability Test of Frail´BESTest in Elderly Institutionalized Frail People
Status: Completed | Type: Observational
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Responsible Party: Principal Investigator, Sandra Calvo Carrión, PhD in Health Sciences, Instituto de Investigación Sanitaria Aragón
Other Study IDs: Validation Frail´BESTest
Record Dates: First submitted 2024-05-27; First posted 2024-06-03 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Frail Elderly Syndrome; Mild Cognitive Impairment
Keywords: Fragility; Mild Cognitive Impairment; Older adult; Institutionalised
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Validation group: This Cross-sectional study consists of five phases. PHASE 1 [T1] Consist on the linguistic validation and it will be carried out the transcultural adaptation of Frail'BESTest in a population sample (named group A), which will be made up of 30 individuals over 60 years of age, community living independently in their houses, cognition preserved, who have a preserved physical functional status, and able to stand up still, without assistive devices for 10s or over (Group A).
  PHASE 2 [T2] consist on reliability. One subgroup (GROUP B and GROUP C) of institutionalized frail aged participants, n=30 with mild cognitive impairment (named group B) and 30 without mild cognitive impairment (named group C) will be tested. We will examine between raters reliability and test-retest reliability.
  PHASE 3 [T3] consisting on construct validity. PHASE 4 [T4] consisting on predictive falls/concurrent validity. PHASE 5 [T4] consisting on predictive decease/concurrent validity.

SUMMARY:
The aging of the global population presents significant social and health challenges. In Aragón, 15% of the population is between 65 and 79 years old, and the over-aging index is 16.6%, higher than the national average. This aging necessitates promoting healthy aging and maintaining functional capacity in advanced ages. Currently, 15% of the Aragonese population is potentially dependent, a figure that rises to 26% among those over 85 years old. The decline in functional capacity is due to auditory, visual, joint, and proprioceptive issues, resulting in increased vulnerability to falls, which are a significant cause of death among the elderly.

The frailty syndrome, although common with aging, is not inevitable and is characterized by the loss of functional capacity and increased risk of falls and hospitalization. To assess this capacity in frail individuals, specific tools like the Mini-Motor Test, the Morton Mobility Index, and the Elderly Mobility Scale exist. The BESTest, developed in 2009, evaluates balance but is time-consuming to administer, leading to the creation of a shorter version, the Mini BESTest. However, both can be limiting for frail individuals.

To address these limitations, the Frail'BESTest was developed, evaluating six balance subsystems and being suitable for frail individuals, making it a valid and sensitive tool in clinical practice. This research project aims to develop tools that identify balance problems in frail individuals with mild cognitive impairment, allowing for specific interventions to reduce the risk of falls.

DETAILED DESCRIPTION:
This is a cross-sectional study consisting of two phases. In the first phase, the linguistic-transcultural validation of the Frail'BESTest will be carried out in a population (which we will call group A), which will be made up of people over 65 years of age who live in a community, who do not present cognitive impairment and whose physical functional state is preserved.

In a second phase of the study, the validity and reliability of the test will be analysed in frail institutionalised people with mild cognitive impairment. For this purpose, frail people with mild cognitive impairment (group B) and frail people with no cognitive impairment (group C), all of them over 65 years of age, will be selected.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be able to maintain 10seconds stand feet apart without assistance The Validity of FRAILBESTest in mild cognitive impairment institutionalized patients will be made of subgroup categories: Frail/Non-frail; Cognition preserved/Mild cognitive impairment patients and Institutionalized patients/community living individuals.
* Frailty will be determine by Fried phenotype Those scoring 3 or more out of 5 will be classify as frail and those scoring 2 or less as non-frail individuals. Mini-Mental State Examination (MMSE) cognition status could be preserved or altered (Score >24-30).
* Community living individuals will be non-frail and cognition should preserved they will be assign to Group A.
* Frail institutionalized individual's (scoring from 24 to 26 at MMSE) will be assign to Group B Frail institutionalized individual's (scoring = or > to 27 at MMSE) will be assign to Group C Non frail Institutionalized individuals with cognition preserved (scoring = or > to 27 at MMSE) will be assign to group D.

Exclusion Criteria:

* Orthopedic unstable conditions
* Moderate or severe cognitive status Score <24 at MMSE
* Inability to understand indications or communicate with testers.
* Sustaining severe cardiac, vascular or respiratory diseases or conditions that contraindicate physical activity
* Presenting a condition for which, in the opinion of the researchers, the evaluation may pose a risk to their health
* Not having autonomy to decide about their voluntary participation in the study

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Group A: Community Living, Non-Frail individuals Cognition preserved (n=30).
  * Group B: Institutionalized Frail with mild cognitive impairment n=240 (divided in two groups, n= 30 and n=210).
  * Group C: Institutionalized Frail without cognitive impairment (n=40).
    * Group B: will be obtained from the users of the residences for the elderly of the Fundación Rey Ardid in Zaragoza: Residencia Rosales and Residencia Juslibol. The recruitment will screen by the physiotherapist working in both residences by a verbal invitation. .
    * Group C: will be obtained from the users of Casa Amparo (Zaragoza) and the residences of the Federico Ozanam Foundation: Perpetuo Socorro (Garrapinillos), CAI-Ozanam Oliver, San Antonio de Padua, Ibercaja Ozanam La Magdalena, Ozanam Santa Isabel and María Auxiliadora (María de Huerva), Hermanitas de los pobres desamparados and the Mazaruba residence in Zaragoza. The authorised health personnel from each of the centres will screen participants and invite them.
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
Frail'BESTest: assesses static, dynamic balance and mobility | Baseline (T0) and 7 days (T1) following baseline.
  6 balance systems are tested, with between 2-6 tests per balance system. The balance systems tested are: A: anticipations, B: reactions, C: locomotion, D: sensorial orientation, E: biomechanical constraints and F: gait symmetry. All tests or criteria are scored dichotomously, with 0 for negative results and 1 for positive results. The highest and best possible score for the Frail'BESTest is 26 and the lowest is 0.
  A. Proactive motor control anticipatory maximum score is 5 and the minimum score is 0 (equivalent to 19%).
  B. Reactive motor control - reactions - maximum score 2 and minimum score 0 (equivalent to 8%).
  C. Locomotion and gait - maximum score 6 and minimum score 0 (equivalent to 23%) D. Static postural control maximum score 3 and minimum score 0 (equivalent to 12%).
  E. Biomechanical restrictions maximum score is 6 and the minimum score is 0 (equivalent to 23%).
  F. Gait symmetry maximum score is 4 and the minimum score is 0 (equivalent to 15%).

SECONDARY OUTCOMES:
The Short Physical Performance Battery (SPPB): assesses functional performance | Baseline (T0) and 7 days (T1) following baseline.
  It is a battery that evaluates functional performance in three functional activities and measures the ability to: 1) maintain three different conditions of static balance for 10 seconds, 2) the time it takes to walk 4 meters and 3) stand up and sit down from a chair 5 consecutive times. Depending on the result, each of the activities is scored from 0 to 4 points, with the maximum possible score being 12 points.
Timed up and Go test (TUG): assess lower limb function | Baseline (T0) and 7 days (T1) following baseline.
  The TUG test (Timed Up and go (TUG) measures the functional mobility of the lower limbs.
  The patient sits on the chair and leans back against the back of the chair; the soles of the feet must be on the floor. On the command "Go"," the patient gets up from the chair (he is not restricted when getting up from the chair, he can use his upper extremities), walks 3 m at a fast, safe pace, turns around, goes back to the chair and sits down. The patient chooses the side on which the turn is to be performed. The timing starts with the instruction "Go" and ends when the patient is seated (buttocks touching the chair).
Dual task cost of naming on gait speed: assesses the ability of executing two tasks (naming and walking) in this case the effect of cognitive task on gait speed. | Baseline (T0) and 7 days (T1) following baseline.
  To calculate dual-task costs of naming on gait, two tests of gait are required. Test 1. Test of single gait at comfortable speed. A test of gait speed assesses an individual's functional mobility. Gait speed is calculated with the time taken to walk 10m distance on level surfaces at their comfortable speed over the entire distance. Examinees will be time once the first foot passes path line; the time is stopped once the first foot enters the 10m path line. Two trials are given. Analysis maximum speed obtained.
  Test 2. Test of gait speed dual task assesses an individual's functional mobility while naming cities from the country patients belong (cognitive activity). The procedure to record time will be the same before. Gait speed will be calculated:
  * Dual task gait speed (m·s-1) = 10m /Time taken to walk 10m naming cities
  * Dual Task Cost of naming on Gait Speed (DTC-GS) will be calculated using the formula:
  * DTC-GS [%] = 100 · (single-task value - dual-task value)/single-task value
Dual task cost of gait on naming: is the ability executing two tasks (naming and walking) and the effect gait activity on naming task. | Baseline (T0) and 7 days (T1) following baseline.
  Quantifies subjects' ability executing two tasks concurrently (naming and walking).
  Test-1: The test of single cognitive task consists of naming towns for 30 seconds. The patient will be seated on a chair. The calculation of the number of towns correctly named per second will be recorded.
  DT Number of towns per seg = number of towns /10m gait dual task (seg) Test-2. Test of gait speed dual task results. While the patient performs the test it will record the time taken to walk 10m distance on level surfaces and the number of cities in the country correctly named, repeated during the 10-meter march.
  The calculation of the number of towns correctly named per second will be recorded Only one trial is given Dual task cost of gait on naming (DTC-N):
  * Dual-task Number of cities per sec = correct number of cities /10m gait dual task (seg)
  * Dual Task Cost of Gait on Naming (DTC-N) will be calculated:
  * DTC-N [%] = 100 · (single-task value - dual-task value)/single-task value
The Mini Balance Evaluation System (MiniBESTest): assess complementary systems that contribute to balance function using static, dynamic balance test and mobility test | Baseline (T0) and 7 days (T1) following baseline.
  The MiniBESTest was developed, and it is having been validated as a shorter version of the original BESTest to assess complementary systems that contribute to balance function. It aims to target and identify 6 different balance control systems so that specific rehabilitation approaches can be designed for different balance deficits. The tests include functional tasks involving several high-level exercises to assess the balance function, which may be even more difficult in case of frailty 1.1. TASKS Mini BESTest is a 14-item test scored on a 3-level ordinal scale (0-2) Total score = 32 points per test directions as we will specify use of both left and right data, thus calculating data based on 32. Assesses dynamic balance, a unidimensional construct and includes 14 items addressing 4 of the 6 sections of the original BESTest: I) Anticipatory postural adjustments II) Reactive postural control III) Sensory orientation IV) Dynamic gait.
Performance Oriented Mobility Assessment (POMA): is also known as Tinetti test. It assesses balance and mobility. | Baseline (T0) and 7 days (T1) following baseline.
  The patient can use any assistive devices during the test. The test comprises two short sections that contain one examining static balance abilities in a chair and then standing, and the other gait. Total POMA consists of 16 items: 9 balance (POMA-B) and 7 gait (POMA-G) items. A 3-point ordinal scale, ranging from 0-2, where highest score indicates independence with each test item.
  2.1. TASKS POMA has 2 sections 1) Assesses balance abilities in a chair and in standing position and 2) Assesses dynamic balance during gait. Total balance score is16 and gait 12; total Test score 28.
  Balance Subscale The patient is to sit in an armless chair and will be asked to rise and stay standing. The patient will then turn 360° and then sit back down. This is to test the patients' balance.
  At gait sub-scale the patient will have to walk a few meters at a normal speed, followed by turning and walking back at a "fast but safe" speed. The patient will then sit back down.
Falls. | 6 months (T2) Following baseline Test.
  Falls are defined as an unexpected event in which the participants come to rest on the ground, floor, or lower level.
  The number of falls, will be obtain from medical history records of nursing homes.
Patient's decease. | 1 year (T3) following baseline.
  Deceases and time to patient's decease will be obtain from medical history records of nursing homes.
Dual task cost of counting backwards on Timed up and Go (TUG): assesses the ability of executing two tasks (counting backwards and performing a mobility test) on the mobility task. | Baseline (T0) and 7 days (T1) following baseline.
  Subjects' ability for executing two tasks concurrently (counting backwards in threes while doing a mobility test named TUG. To calculate dual-task costs of counting backwards on TUG The test is conducted single (TUG) and dual tasking, counting backwards in three (TUG-3). Two trials will be record for each condition and the best them will use for further analysis.
  Test-1-TUG. The patient sits with his/her back against the chair; the soles of feet must be on the ground. On the command "Go," the patient rises from the chair, walks at fast pace safe manner for 3m, turns, walks back to the chair and sits down.
  Test-2-TUG-3. Records time needed to complete TUG test while counting backward by threes. Different starting numbers will be use for the counting tasks.
  Dual Task Cost of counting backwards in threes on TUG (DTC-3-TUG) will be calculate using the formula:
  DTC-3-TUG [%] = 100 · ((single-task value - dual-task value)/single-task value)).

CONTACTS AND LOCATIONS:
Overall Officials: María del Pilar Domínguez Oliván, PhD, Principal Investigator — Universidad de Zaragoza
Locations (1):
- Universidad de Zaragoza, Zaragoza, Zaragoza, Spain